CLINICAL TRIAL: NCT03108586
Title: Caries Associated With Restorations or Sialants Cognition and Identification in Adults
Brief Title: Caries Cognition and Identification in Adults
Acronym: CaCIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: UFPEL- PPGO 0020
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Secondary Caries
Keywords: restorations; diagnosis; secondary caries; treatment decision
MeSH Terms: conditions — Disease | interventions — Dental Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, clinical operators responsible for dental treatment, and the examiner who will assess the outcomes will be blind to the allocation group of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FDI - tradional group (Active Comparator): Diagnosis and dental treatment decision based on the criteria of the International Dental Federation (FDI).
  Interventions: Procedure: Dental treatment
- CARS - conservative group (Experimental): Diagnosis and dental treatment decision according to CARS (Caries Associated with Restorations or Sealants) detection criteria.
  Interventions: Procedure: Dental treatment

INTERVENTIONS:
Procedure: Dental treatment — Dental treatment of all dental needs present in adults related or not to the dental caries
  Arms: FDI - tradional group
Procedure: Dental treatment — Dental treatment of all dental needs present in adults related or not to the dental caries
  Arms: CARS - conservative group

SUMMARY:
This study will evaluate the effect of the International Dental Federation (FDI) criteria, compared to CARS (Caries Associated with Restorations or Sealants) detection criteria for evaluation of caries lesions around restorations in permanent teeth, in the outcomes related to oral health of adults, in a randomized clinical trial.

DETAILED DESCRIPTION:
The study will consist of a randomised controlled trial of two parallel groups. One group will correspond to adults who will receive the diagnosis and indication of treatment according to the standard criteria, following the FDI criteria to classify the restorations marginal conditions and the presence of secondary caries (traditional group). And the other group will receive a diagnosis and treatment decision according to a minimal intervention approach, using as reference the detection criteria "Caries Associated with Restorations or Sealants" (CARS) - ICCMS (International Caries Classification and Management System) - conservative group). Patient evaluations will be performed yearly after 12 months. The primary outcome will be the number of surfaces restored with the need for new interventions. Secondary outcomes will be the impact of oral health on quality of life and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking dental treatment at the School of Dentistry;
* Age between 18 and 60 years;
* Patients who present at least one restoration of composite resin or amalgam to posterior and/or anterior teeth.

Exclusion Criteria:

* Patients who refuse to participate in the research;
* Patients included in other surveys that involve restorations or are in systematic attendance at another clinic or service;
* Patients who present systemic conditions or chronic diseases that require differentiated care and follow-up - these will be referred to the specific services available at the Faculty of Dentistry;
* Patients who reside in other locations and who can not return for periodic follow-up of the interventions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in number of surfaces restored requiring new intervention | 12 months, 24 months
  The primary endpoint will be the number of surfaces restored requiring intervention, which is composed of the sum of components with different levels of severity: number of surfaces with new caries lesions, number of surfaces restored in need of repair, replacement, teeth with episodes of pain, teeth requiring endodontic treatment or extraction.

SECONDARY OUTCOMES:
Impact of intervention on quality of life measured by a validated questionnaire - OHIP-14 (Oral Health Impact Profile-14) | 12 months, 24 months
Cost-effectiveness measured by a scale | 12 months, 24 months
  Effectiveness will be measured through the number of restored surfaces without intervention. The cost-effectiveness ratio will be expressed by the cost ratio of the FDI and CARS criteria and effectiveness (number of surfaces without the need for new interventions)

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano Cenci, PhD, Principal Investigator — Federal University of Pelotas
Locations (2):
- Brazil (2):
  - Federal University of Pelotas, Pelotas, Rio Grande do Sul
  - School of Dentistry - Federal University of Pelotas, Pelotas, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Signori C, Moro BLP, Uehara JLS, Romero VHD, de Oliveira EF, Braga MM, Mendes FM, Cenci MS; CaCIA Collaborative Group. Study protocol for a diagnostic randomized clinical trial to evaluate the effect of the use of two clinical criteria in the assessment of caries lesions around restorations in adults: the Caries Cognition and Identification in Adults (CaCIA) trial. BMC Oral Health. 2020 Nov 10;20(1):317. doi: 10.1186/s12903-020-01307-z. PMID 33172449
- [Result] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Result] Brouwer F, Askar H, Paris S, Schwendicke F. Detecting Secondary Caries Lesions: A Systematic Review and Meta-analysis. J Dent Res. 2016 Feb;95(2):143-51. doi: 10.1177/0022034515611041. Epub 2015 Oct 13. PMID 26464398